CLINICAL TRIAL: NCT01595620
Title: Cannabinoid Modulation of Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 1005006859
Record Dates: First submitted 2012-04-25; First posted 2012-05-10 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Pain
Keywords: Cannabis; THC; Pain
MeSH Terms: conditions — Pain; Marijuana Abuse | interventions — Electricity; Capsaicin; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- THC 0.01 mg/kg (Active Comparator)
  Interventions: Other: Thermal; Other: Electrical; Other: Capsaicin; Drug: THC
- Placebo (Placebo Comparator)
  Interventions: Other: Thermal; Other: Electrical; Other: Capsaicin; Drug: Placebo
- THC 0.03 mg/kg (Active Comparator)
  Interventions: Other: Thermal; Other: Electrical; Other: Capsaicin; Drug: THC

INTERVENTIONS:
Other: Thermal — Thermal sensation/pain testing
Other: Electrical — Electrical sensation/pain testing
Other: Capsaicin — Intradermal Capsaicin
Drug: THC — Active THC (0.01 mg/kg) administered over 10 minutes
  Other Names: Delta-9-tetrahydrocannabinol
  Arms: THC 0.01 mg/kg
Drug: THC — Active THC (0.03 mg/kg) administered over 10 minutes
  Other Names: Delta-9-tetrahydrocannabinol
  Arms: THC 0.03 mg/kg
Drug: Placebo — Control: small amount of alcohol with no THC, administered over 10 minutes
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effects of cannabinoids on pain response using a variety of human experimental pain models.

ELIGIBILITY:
Inclusion Criteria:

* At least one lifetime exposure to cannabis
* Acceptable Birth Control methods for females

Exclusion Criteria:

* Cannabis naive
* Medical or psychiatric contraindications
* Analgesic medication
* Previous sensitivity to THC or cannabis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11-09 (Actual); Primary Completion 2012-04-19 (Actual); Study Completion 2012-04-19 (Actual)

PRIMARY OUTCOMES:
Capsaicin-induced hyperalgesia | On each test day at baseline (-30), peak (+20) and post (+120) drug administration

SECONDARY OUTCOMES:
Pain Measures | On each test day at baseline (-30), peak (+20) and post (+120) drug administration
Non-pain subjective responses | On each test day at baseline (-30), peak (+20) and post (+120) drug administration
Cognitive subjective responses | On each test day at baseline (-30), peak (+20) and post (+120) drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States